CLINICAL TRIAL: NCT02752555
Title: Investigating the Effect of Modifiable Lifestyle Factors in Severe Oligoasthenotertozoospermic Men Combined With Antioxidant Treatment Prior ICSI
Brief Title: Severe Male Factor Infertility Management
Acronym: OAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Salah Elbashir, Assisting lecturer of Urology, Benha University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00287597
Record Dates: First submitted 2016-04-23; First posted 2016-04-27 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Oligoasthenoteratozoospermia
Keywords: Oligoasthenoteratozoospermia; Male factor managment; Intacytoplasmic sperm injection
MeSH Terms: conditions — Oligospermia | interventions — Antioxidants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Antioxidant group (No Intervention): In the control group, all patients will go a double-blind therapy of a three-months period of treatment with oral carnitine (2g daily). After this period, all patients will undergo conventional intacytoplasmic sperm injection (ICSI).
- Antioxidant+modifiable lifestyle factors (Experimental): In the study group, all patients underwent a double-blind therapy of a six-month period of treatment with oral carnitine (2g daily) combined with modifiable lifestyle factors. Patients were requested to follow a healthy standard diet, avoid excessive heat exposure, avoid or minimize exposure to pollutants, and stop smoking, coffee, alcohol, and drugs uptake.After this period, all patients will undergo conventional ICSI.
  Interventions: Other: Antioxidant (l-cratinine) + modifiable lifestyle factors

INTERVENTIONS:
Other: Antioxidant (l-cratinine) + modifiable lifestyle factors — All participants were subjected to the same three-month period treatment protocol, which included 1) antioxidant treatment with L-Carnitine (2g daily); 2) frequent ejaculation every 2 days; and 3) minimizing adverse lifestyle factors.
  Arms: Antioxidant+modifiable lifestyle factors

SUMMARY:
This study is the first to evaluate the effect of oral supplementation with antioxidants combined with lifestyle modification for severe male factor partner of couples undergoing ICSI.

DETAILED DESCRIPTION:
Patients underwent a therapy of a three-month period of treatment with either oral L-carnitine only (2g daily) or oral carnitine (2g daily) combined with modifiable lifestyle factors.

ELIGIBILITY:
Inclusion Criteria:

* Long protocol for ovulation
* Oligoasthenoteratozoospermic male partner ( (count < 0.5 million/ml, Motility=< 40% Progressive motility =<10 %, Abnormal forms >99%).
* Fresh semen samples.

Exclusion Criteria:

* Day 3 embryo transfer
* Incomplete ICSI cycles
* Endometrial thickness> 7mm

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | two weeks
Implantation rate | one month

CONTACTS AND LOCATIONS:
Overall Officials: Salah Elbashir, Study Director — Department of Urology, Benha university, Egypt
Locations (3):
- Egypt (3):
  - Dar Almaraa fertility and gynacology center, Cairo
  - Elite fertility care center, Cairo
  - Nile badrawi Hospital, Cairo

IPD SHARING:
Plan to Share IPD: Yes
Publishing a manuscript

REFERENCES:
- [Background] Tremellen K, Miari G, Froiland D, Thompson J. A randomised control trial examining the effect of an antioxidant (Menevit) on pregnancy outcome during IVF-ICSI treatment. Aust N Z J Obstet Gynaecol. 2007 Jun;47(3):216-21. doi: 10.1111/j.1479-828X.2007.00723.x. PMID 17550489